CLINICAL TRIAL: NCT02393911
Title: Dysbiosis in the Vaginal Microbiota May be Associated With the Development of Localized Provoked Vulvodynia (LPV)
Brief Title: Dysbiosis in Localized Provoked Vulvodynia (LPV)
Acronym: DMLPV
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Prof. Jacob Bornstein, Principal Investigator, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 0146-14-NHR
Record Dates: First submitted 2015-01-27; First posted 2015-03-20 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Vulvodynia; Vulvar Vestibulitis
Keywords: vestibulitis; microbiome
MeSH Terms: conditions — Vulvodynia; Vulvar Vestibulitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Study A - with diet (Active Comparator): Patients with LPV, treated by Low Oxalate Diet for three months.
  Interventions: Dietary Supplement: Low Oxalate Diet
- Study B- no diet (Active Comparator): Patients with LPV, not treated by Low Oxalate Diet for three months.
  Interventions: Dietary Supplement: Low Oxalate Diet
- Control (Active Comparator): Healthy women without LPV, not treated by Low Oxalate Diet
  Interventions: Dietary Supplement: Low Oxalate Diet

INTERVENTIONS:
Dietary Supplement: Low Oxalate Diet — Low oxalate diet is a diet where products with oxalate will be eliminated, such as: tomatoes, berries, coffee, nuts

SUMMARY:
Currently, the pathogenesis of Localized Provoked Vulvodynia (LPV) has not been elucidated. Few observations may point to involvement of the microbiome: the association of LPV with preceding chronic recurrent candidiasis, and the reports of the beneficial effect of a diet avoiding oxalate on Vulvodynia.

Studies in the new field of microbiome research focus on the composition of overall microorganisms in our body and their impacts on our health. Changes in the composition of the vaginal microbiota (dysbiosis) have been linked with different health and disease states. We have also shown recently that women can be divided into 2 groups according to the composition of their vaginal microbiome.

The proposed study will compare the vaginal microbiome of women with severe LPV, not treated by diet and otherwise healthy, to women without LPV (we will also compare our results to the NIH HMP data). Vaginal pH and date of menstrual cycle will be checked. We propose that dysbiosis in the vaginal microbiota may trigger the development of LPV.

DETAILED DESCRIPTION:
Vulvodynia - vulvar pain. The exact etiology has not been elucidated yet, and therapy is often unsatisfactory. Two main types of Vulvodynia exist, with the far more common type being Localized provoked vulvodynia (LPV), also known as Vestibulodynia, and in the past - Vestibulitis. This study will concentrate on this common disorder which affects young women, whose quality of life deteriorate significantly by the inability to experience vaginal sex.

The vaginal microbiome The new field of microbiome research focuses on the composition of overall microorganisms in the human body and their impacts on our human health. Amazingly, the number of microbial cells within our body is 10 times greater than the sum of all our human somatic and germ cells, and they carry 150 times more genetic information than our own. Changes in the composition of the vaginal microbiota (dysbiosis) have been linked with different health and disease states.

The vagina is colonized with around 108-109 bacteria/mL vaginal fluid which is comparable to the small intestine. Recently, the NIH Human Microbiome Project characterized the bacterial communities across the human body and found that the vagina harbors low complexity bacterial communities. These communities had the lowest alpha diversity (within sample diversity) among the different body sites and low beta diversity (between sample diversity) at the genus level. This diversity was high at the species level due to distinct Lactobacillus spp. The communities were sampled at the sub sites that included the posterior fornix, mid vagina and the vaginal introitus. There was little distinction between the three sites hence we will focus on posterior fornix. The vaginal communities of healthy women, have also been repeatedly observed to occupy one of five states, four dominated by Lactobacillus spp. and one by higher overall microbial diversity. Shifts between the community structures within individuals (dysbiosis) are associated with disease states so it would be interesting to study whether women with LPV belong to a different enterotype than healthy women.

The vaginal microbial communities have been shown to change during different stages in a woman's life and to influence pregnancy. As early as 1930, Cruickshank and Baird described changes in the vaginal bacterial communities that occurred between the 5th and 7th month of pregnancy.

In 2010 a study was undertaken among Amerindian women to examine the microbial vaginal signature at term in relation to delivery mode (n=9). Variability in vaginal taxa was noted between subjects particularly for Lactobacillus species. Metagenomic analysis of the vaginal microbiome in a cross-sectional study of 24 healthy pregnant women and 60 non-pregnant controls at three vaginal sites (introitus, posterior fornix and midvagina) found the richness and diversity of the vaginal microbiome to be reduced in pregnancy in ways that did not appear to be driven by BMI, race or ethnicity . As pregnancy progressed and as proximity to the uterus increased, less diversity and richness were noted. Lactobacillus species were enriched in pregnancy, which the authors postulated may be biologically significant as lactic acid bacteria produce bacteriocins that may reduce the risk of ascending infections. It has also been proposed that the vaginal microbiota has the potential to influence the conception process by influencing the local production of proinflammatory cytokines which in turn impact the survival rate and motility of sperm cells.

The vaginal microbiome and Vulvodynia Several microorganisms have been discussed for presumed role in LPV development: LPV is frequently associated with preceding chronic recurrent candidiasis, LPV may be produced in a mouse model by repeated vulvovaginal fungal infection, the difficulty in treating women with concomitant LPV and candidiasis (complicated LPV), the reports of the beneficial effect of treatment with combined antibiotics, aimed at eradicating H. pylori peptic condition (although H. pylori has not been detected in LPV tissues).

Indirect evidence of the role of the microbiome with the development of LPV may be deduced from the beneficial effect (14.3 - 50%), reported by some authors, of a diet avoiding oxalate and rich in Calcium citrate, on LPV. As women with LPV consume more oxalate - although not significantly, we suspect that the variability in response rate may be due to the indirect effect of the diet - through changes in the microbiome, which may be affecting LPV severity. In addition, the adverse effect of oral contraceptive pills (OCP) in increasing LPV symptoms; OCP tend to change the composition of the vaginal microbiota, consequent to their effect of thinning and dehydrating the vaginal mucosa. These finding prompt us to further inquire the possible association of vaginal microbiome dysbiosis and the development of LPV.

Objective:

The proposed study will first compare the vaginal microbiome of women with severe LPV, not treated by diet and otherwise healthy, to women without LPV (we will also compare our results to the NIH HMP data). At the second stage we will characterize the effect of a three-month low oxalate diet on the vaginal microbiota of women with LPV and on the outcome compared to a group of patients with LPV not treated by diet. Vaginal pH and date of menstrual cycle will be checked. We propose that dysbiosis in the vaginal microbiota may trigger the development of LPV.

Vulvodynia subtype:

* The research will study women with localized provoked Vulvodynia
* Only secondary type of LPV will be included.
* LPV diagnosis will be based on documenting first two Friedrich's criteria for vulva vestibulits syndrome: patient's complaint of entry dyspareunia, a positive Q-tip test.
* Only women suffering from levels II or III dyspareunia according to Marinoff : Level II is where the pain prevents intercourse from taking place on most occasions; and Level III where pain results in total apareunia.

Methods/Protocol This will be a double blind, prospective study comparing the microbiome of women with severe LPV to women without LPV, and to compare the effect of consuming the low oxalate diet with calcium citrate supplements for one month on the microbiome of women with LPV.

The local Institutional Review Board approval has been requested. Every woman participating in the study will sign an informed consent prior to enrollment.

Study group

The study group will consist of 35 women:

* Meeting first two Friedrich's criteria for vulva vestibulitis syndrome
* Diagnosed by a gynecological examination with Localized Provoked Vulvodynia
* Diagnosed with a Level II or III degree of the syndrome according to Marinoff Control group
* The control group will consist of 35 consecutive women who are referred to the departments of the co-investigators. Presentation of LPV is an exclusion criterion.

Materials and Methods:

Prior to enrollment, the women will be questioned about possible inclusion and exclusion criteria, and fill in the ISSVD Vulvodynia questionnaire.

Women found suitable for the study will undergo a Q-tip test to confirm the diagnosis of Vestibulodynia. Women of the LPV group will be instructed to consume a "low oxalate diet" with calcium citrate supplements, as recommended by Solomons et al for the duration of at least one month, to assess its impact on the vaginal microbiome.

Clinical pain scores and vulvar sensitivity by Q-tip test will be repeated after one month and compared to the clinical pain scores at the beginning of the study. Subjective evaluation will be carried out by comparing personal data from questionnaires filled in at enrollment and one month later.

Clinical evaluation will be performed by an experienced vulvar expert, using the pain intensity scale (The 11 points (0-10) pain intensity numerical rating scale-PI-NRS), in seven foci throughout the vestibule (the Q-tip test) and by comparing patients' responses to questionnaires evaluating pain during intercourse or other activities (riding a bicycle/horse), before and after diet.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women, aged 18-50 years, meet Friedrich's first two criteria for vulvar Vestibulitis syndrome, suffer from levels II or III dyspareunia according to Marinoff

Exclusion Criteria:

* Women suffering from generalized Vulvodynia (constant vulvar pain - unrelated to provocation), pregnant or lactating. Women will also be excluded from the study if they were have any medical condition, acute or chronic, or anticipated not being available for the one month follow up visit, have received antibiotics during the month preceding the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Change in vaginal microbiome composition of women with localized provoked vulvodynia following three months of low oxalate diet | Within one week after three months of low oxalate diet
  The microbiome components will be examined before and after the diet by characterization of the genomic components of the bacterial communities

SECONDARY OUTCOMES:
Level of dyspareunia following three months of low oxalate diet in women with localized provoked vulvodynia | Within one week after three months of low oxalate diet
  The level of vestibular tenderness will be examined before and after the diet

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Bornstein, MD, Principal Investigator — Western Galilee Hospital

REFERENCES:
- [Derived] Awad-Igbaria Y, Palzur E, Nasser M, Vieira-Baptista P, Bornstein J. Changes in the Vaginal Microbiota of Women With Secondary Localized Provoked Vulvodynia. J Low Genit Tract Dis. 2022 Oct 1;26(4):339-344. doi: 10.1097/LGT.0000000000000689. Epub 2022 Aug 6. PMID 35943448